CLINICAL TRIAL: NCT04788875
Title: Small Bite Technique Versus Standardised Large Bites Technique in Closure of Midline Laparotomies: Randomised Control Trial.
Brief Title: Small Bite Technique Versus Standardised Large Bites Technique in Closure of Midline Laparotomies.
Acronym: SBT-CML
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Nasser Mohamed Amer, Assistant professor of General Surgery in Imam Abdulrahman bin Faisal University, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SBT-CML
Record Dates: First submitted 2021-02-09; First posted 2021-03-09 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Incision, Surgical; Suture, Complication; Incisional Hernia
MeSH Terms: conditions — Surgical Wound; Incisional Hernia

STUDY DESIGN:
Intervention Model Description: 2 Arms Arm1) Closure of laparotomy by small bites technique using PDS 2.0 Arm2) Closure of laparotomy by standardised large bites technique
  This research will include all patients who will had laparotomy through a midline incision according to our inclusion criteria, they will be randomised using computer generated numbers by using (Random.org), to either closure by small bites technique using PDS 2.0 or standardised large bites technique.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded. (patients and research recruiter)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small Bite Technique Group (Active Comparator): closure of laparotomy by small bites technique using PDS 2.0
  Interventions: Procedure: Small bite suturing Technique
- Standardised Large Bites Technique Group (Other): usual practice closure of laparotomy by standardised large bites technique using PDS 2.0
  Interventions: Procedure: Standardised Large Bites Technique

INTERVENTIONS:
Procedure: Small bite suturing Technique — Small bite suturing technique with PDS 2.0
  Arms: Small Bite Technique Group
Procedure: Standardised Large Bites Technique — Standardised large bite suturing technique with PDS 2.0
  Arms: Standardised Large Bites Technique Group

SUMMARY:
In the attempt to gain quick and complete access to the abdominal regions with the least damage to the nerves and the vascular structures, surgeons use the median laparotomy more frequently. However, postoperative complications such as incisional hernia continue to be the known leading complications after median laparotomy. The reported cases to range from 2 to 20%. Higher cases have also been reported with up to 35% in the absence and aortic patients. Recent statistics have showed that small tissue bites prevent incisional hernia can occur in the aponeurosis. This technique is more effective than the commonly used process, which involves large edges of mass closure. In this study investigators aim to compare small bites sutures in closure of laparotomy incision and standardized large bites sutures, and its affect in reducing the incidence of incisional hernia postoperative along with the surgical site infection.

the investigators hypothesize that the small bites technique will result in a significant reduction of the incidence of incisional hernia and optimize the surgical site infection in major surgeries which may lead to a reduced morbidity and a better quality of life for patients and a significant reduction of costs.

DETAILED DESCRIPTION:
Incisional hernia carries with life-threatening conditions such as the incarceration of bowel strangulation. However, incisional hernia remains the most common complication after median laparotomy, with reported incidences varying between 2-20%. Even higher incidences up to 30-35% have been reported in obese and aortic aneurysm patients. Incisional hernia also causes life impairment and discomfort. Median laparotomy and the incisional hernia have been under investigation for quite some time, and information about patients' risk factors and suture materials has been identified. However, the risk factors associated with suture techniques are not yet thoroughly investigated. Many clinical tests and analyses have concluded that a mass closure technique involving a simple running suture is the most effective way to prevent incisional hernia and close a midline incision. The method is also easy and fast to perform compared to other layered methods involving interrupted sutures. Use of natural materials that are thin resorbable materials decreases the occurrence of the incisional hernial and lower the intensity of preoperative pain and wound infections compared to the use of suture materials that are non-resorbable.

In this study the investigators aim to compare the small bites technique with a standardised large bites technique:

* Primary outcome:

  1. Incidence of Incisional Hernia postoperative.
  2. Pain scale.
* Secondary outcome:

  1. Quality of life, recovery, return to usual activity.
  2. Surgical site infection
  3. Time for closure.

     Study Design:
* Randomized Control Trial, Double blinded.

Study area\ sitting :

- The study will be conducted in King Fahad University Hospital, Khobar, Eastern Province, Saudi Arabia.

Sample size:

108 patients

Number of Arms (allocation):

2 Arms Arm1) Closure of laparotomy by small bites technique using PDS 2.0. Arm 2) Standardised large bites technique.

Randomisation technique:

Random.org

Blinding technique:

Double blinded. (patients and research recruiter) Follow up period: 6 months then 1 year, follow up by US.

Outcome expected to measure:

Study Subjects :

* Inclusion criteria:

  1. Laparotomy through a midline incision
  2. Age more than 18
  3. BMI < 40
* Exclusion criteria:

  1. Previous incisional hernia or fascial dehiscence with secondary healing after a midline incision.
  2. Abdominal surgery through a midline incision within the last three months.
  3. Pregnancy.
  4. Patient on steroids and with genetic anomalies.
  5. Malignancy patients, next exposed to radiation therapy.

Data Collection methods, instruments used, and measurements:

This research will include all patients who will had laparotomy through a midline incision according to our inclusion criteria, they will be randomised using computer generated numbers by using (Random.org), to either closure by small bites technique using PDS 2.0 or standardised large bites technique. The surgery will be done by either a consultant or a specialist following standard steps. A data sheet of each patient regarding their demographic, operation data, and postoperative recovery (pain, early mobilizing, wound healing, surgical site infection, retain to usual activity), then all patients will be followed for 6 month and 1 year postoperative by US, the endpoint is discovering of incisional hernia or not for 1 year follow up.

Data Management and analysis plan:

* SPSS will be used for data analysis.
* Summary statistic will be obtained as frequency, and percentage for qualitative data, and means, medians and standard deviations from continuous variables.
* Chi square test will be used to examine the significant difference of hernia rate between the two study group.
* T test will be used to examine the difference in the mean of pain post-operative between the two study group.

Ethical Considerations:

* Our study does not have any physical, psychological, social, legal, economic risk.
* The study will be reviewed by IRB, ethics committee; then the approval will be obtained.
* Written approval will be obtained from the patients prior to the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Laparotomy through a midline incision
2. Age more than 18
3. BMI < 40

Exclusion Criteria:

1. Previous incisional hernia or fascial dehiscence with secondary healing after a midline incision.
2. Abdominal surgery through a midline incision within the last three months.
3. Pregnancy.
4. Patient on steroids and with genetic anomalies.
5. Malignancy patients, next exposed to radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Incisional Hernia postoperative | Follow up on 6 month postoperative.
  Incidence of Incisional Hernia postoperative, will be assessed by using Ultra Sound.
Incidence of Incisional Hernia postoperative | Follow up on 1 year postoperative.
  Incidence of Incisional Hernia postoperative, will be assessed by using Ultra Sound.
Assessment of pain severity postoperative by pain scale | Day 1 postoperative
  Assessment of pain scale post operative, lower score mean a better outcome.
Assessment of pain severity postoperative by pain scale | Day 2 postoperative
  Assessment of pain scale post operative, lower score mean a better outcome.
Assessment of pain severity postoperative by pain scale | Day 3 postoperative
  Assessment of pain scale post operative, lower score mean a better outcome.
Assessment of pain severity postoperative by pain scale | Day 4 postoperative
  Assessment of pain scale post operative, lower score mean a better outcome.
Assessment of pain severity postoperative by pain scale | Day 5 postoperative
  Assessment of pain scale post operative, lower score mean a better outcome.
Assessment of pain severity postoperative by pain scale | Day 6 postoperative
  Assessment of pain scale post operative, lower score mean a better outcome.
Assessment of pain severity postoperative by pain scale | Day 7 postoperative
  Assessment of pain scale post operative, lower score mean a better outcome.
Assessment of pain severity postoperative by pain scale | Day 8 postoperative
  Assessment of pain scale post operative, lower score mean a better outcome.
Assessment of pain severity postoperative by pain scale | Day 9 postoperative
  Assessment of pain scale post operative, lower score mean a better outcome.
Assessment of pain severity postoperative by pain scale | Day 10 postoperative
  Assessment of pain scale post operative, lower score mean a better outcome.
Assessment of pain severity postoperative by pain scale | Day 11 postoperative
  Assessment of pain scale post operative, lower score mean a better outcome.
Assessment of pain severity postoperative by pain scale | Day 12 postoperative
  Assessment of pain scale post operative, lower score mean a better outcome.
Assessment of pain severity postoperative by pain scale | Day 13 postoperative
  Assessment of pain scale post operative, lower score mean a better outcome.
Assessment of pain severity postoperative by pain scale | Day 14 postoperative
  Assessment of pain scale post operative, lower score mean a better outcome.

SECONDARY OUTCOMES:
Assessment of early mobilisation | Postoperative period, assessment in day1.
  When the patient started to mobilise? assessed by monitoring the patients postoperative and record when he started to mobilise.
Assessment of early mobilisation | Postoperative period, assessment in day2.
  When the patient started to mobilise? assessed by monitoring the patients postoperative and record when he started to mobilise.
Assessment of early mobilisation | Postoperative period, assessment in day3.
  When the patient started to mobilise? assessed by monitoring the patients postoperative and record when he started to mobilise.
Retain to work (how many days between surgery and patient back to his work) | up to 6 weeks, postoperative period from discharge until day patient back to work.
  When the patient back to his work or usual activity? assessed by monitoring the patients postoperative and record when he started to work again.
Surgical site infection of the wound postoperative | day 1 postoprtaive.
  Surgical site infection of the wound postoperative, if there is any sign of surgical site infection, itching, discharge, redness, fever, collection.
Surgical site infection of the wound postoperative | day 2 postoprtaive.
  Surgical site infection of the wound postoperative, if there is any sign of surgical site infection, itching, discharge, redness, fever, collection.
Surgical site infection of the wound postoperative | day 3 postoprtaive.
  Surgical site infection of the wound postoperative, if there is any sign of surgical site infection, itching, discharge, redness, fever, collection.
Surgical site infection of the wound postoperative | day 4 postoprtaive.
  Surgical site infection of the wound postoperative, if there is any sign of surgical site infection, itching, discharge, redness, fever, collection.
Surgical site infection of the wound postoperative | day 5 postoprtaive.
  Surgical site infection of the wound postoperative, if there is any sign of surgical site infection, itching, discharge, redness, fever, collection.
Surgical site infection of the wound postoperative | day 6 postoprtaive.
  Surgical site infection of the wound postoperative, if there is any sign of surgical site infection, itching, discharge, redness, fever, collection.
Surgical site infection of the wound postoperative | day 7 postoprtaive.
  Surgical site infection of the wound postoperative, if there is any sign of surgical site infection, itching, discharge, redness, fever, collection.
Surgical site infection of the wound postoperative | day 8 postoprtaive.
  Surgical site infection of the wound postoperative, if there is any sign of surgical site infection, itching, discharge, redness, fever, collection.
Surgical site infection of the wound postoperative | day 9 postoprtaive.
  Surgical site infection of the wound postoperative, if there is any sign of surgical site infection, itching, discharge, redness, fever, collection.
Surgical site infection of the wound postoperative | day 10 postoprtaive.
  Surgical site infection of the wound postoperative, if there is any sign of surgical site infection, itching, discharge, redness, fever, collection.
Surgical site infection of the wound postoperative | day 11 postoprtaive.
  Surgical site infection of the wound postoperative, if there is any sign of surgical site infection, itching, discharge, redness, fever, collection.
Surgical site infection of the wound postoperative | day 12 postoprtaive.
  Surgical site infection of the wound postoperative, if there is any sign of surgical site infection, itching, discharge, redness, fever, collection.
Surgical site infection of the wound postoperative | day 13 postoprtaive.
  Surgical site infection of the wound postoperative, if there is any sign of surgical site infection, itching, discharge, redness, fever, collection.
Surgical site infection of the wound postoperative | day 14 postoprtaive.
  Surgical site infection of the wound postoperative, if there is any sign of surgical site infection, itching, discharge, redness, fever, collection.
Time taken in closure of laparotomy incision (in minutes) | intraoperative (through the closure of the laparotomy incision inside the operation room, suturing time (start to end) in minutes . (how many minutes surgeon took in suturing the incision))
  Time taken for closure of the laparotomy incision, there will be timer, started from the beginning of suturing the laparotomy incision till the end. (in minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser M Amer, Principal Investigator — Imam Abdulrahman Bin Faisal University